CLINICAL TRIAL: NCT05144893
Title: CPO Pilot: Brief Virtual Mindfulness Based Group Intervention with Social Support
Brief Title: Brief Virtual Mindfulness-based Group Intervention with Social Support for Perinatal Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Oregon (Other)
Responsible Party: Principal Investigator, Kristen Mackiewicz Seghete, Assistant Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00022406
Record Dates: First submitted 2021-11-08; First posted 2021-12-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-04

CONDITIONS: Substance Use; Pregnancy Related; Mental Health
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Mindfullness-Based Support Group (Experimental): The virtual mindfulness-based intervention with social support groups will meet once a week for 4 weeks, each session will be 60 minutes. Each group will have 3-8 participants. The groups will be closed, meaning the same group of participants meet with the same instructor (unless a backup instructor is needed due to unavoidable reasons). Groups will be completed using the video conferencing application.
  Interventions: Behavioral: Virtual Mindfullness-Based Intervention

INTERVENTIONS:
Behavioral: Virtual Mindfullness-Based Intervention — Virtual administration of the social support components of an adapted 4-week Mindfulness Based Cognitive Therapy for Postpartum Depression (MBCT-PD) intervention. Each session includes a review of assigned online mindfulness practice and barriers to practice, other homework if also assigned, psychoeducation, and mindfulness practices relevant to the session's theme.

SUMMARY:
This is a feasibility and acceptability study for 4- week virtual mindfulness-based intervention with social support for perinatal individuals at higher risk for substance use. This study builds on the longitudinal collection of questionnaire data from pregnant and postpartum people during the COVID-19 pandemic. Each closed virtual support group will meet weekly for 4 weeks using a video conference platform. Groups will be focused on grounding, thinking patterns, self-compassion and self-care. This approach will foster increase awareness of wellbeing as well as social support between group participants. Primary outcomes include the feasibility and acceptability of this group-based intervention for perinatal individuals.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant
* Have a single gestation pregnancy
* Fluently speak English
* A history of significant substance use or currently in treatment for a substance use disorder.

Exclusion Criteria:

* Inability to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Interest | at 1 week
  the number of individuals interested in participation.
Feasibility - Attendance | up to 2 months
  the number of individuals who attend group and the average number of groups attended.
Acceptability | up to 2 months
  Acceptability will be assessed using the Customer Satisfaction Questionnaires (CSQ-8). Scores range from 8-32 with higher scores indicating higher satisfaction.

SECONDARY OUTCOMES:
Pregnancy-specific stress | up to 2 months
  Pregnancy-specific stress will be measured using and the Prenatal Distress Questionnaire (PDQ). Scores range from 0 to 46 with higher scores indicating higher distress.
Psychological Distress | up to 2 months
  Overall psychological distress will be measured using the Center for Epidemiological Studies Depression - Revised (CESD-R). Scores range from 0 to 60 with higher scores indicating more severe depressive symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Mackiewicz Seghete, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results of this study will be shared with proper approval.
Supporting Information: SAP
Time Frame: 12 months after final data collectins is concluded through 2 years after publications.
Access Criteria: The Principal Investigator (PI) will review requests for individual participant data (IPD). IPD will be provided with appropriate Institutional Review Board approval or determination. IPD may be provided to investigators associated with a university or reputable research institution with an associated Institutional Review Board (IRB). De-identified IPD will be provided through a secure sharing mechanism.